CLINICAL TRIAL: NCT01133717
Title: Spatial and Temporal Response of Cerebrovascular Response in OSA
Brief Title: Cerebrovascular Reactivity in Obstructive Sleep Apnea (OSA) Subjects
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 09-0831-BE
Record Dates: First submitted 2010-05-20; First posted 2010-05-31 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2010-10

CONDITIONS: Sleep Apnea
Keywords: Sleep Apnea; Cerebrovascular Reactivity
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control without Sleep Apnea
- Subjects with Sleep Apnea

SUMMARY:
Obstructive sleep apnea (OSA) is a prevalent sleep breathing disorder in the general population in which recurrent collapse of the upper airway occurs during sleep. OSA is more prevalent in subjects with stroke and is associated with a 3 fold increased risk of stroke. This makes it a serious public health problem. Approximately 50% of subjects with OSA are asymptomatic and are often only detected following investigation for the cause of heart disease or a stroke. In subjects who are treated for OSA many are intolerant or poorly compliant with treatment. Therefore, the identification of those subjects with OSA most at risk of adverse consequences such as stroke is important, so that treatment compliance can be improved.

Therfore, the investigators want to determine if compared to subjects without OSA, subjects with OSA have evidence of increased stroke risk by assessment of changes in cerebral blood flow (cerebrovascular reactivity) as measured on Doppler ultrasound of the middle cerebral artery (TCD) and blood oxygen level-dependent magnetic resonance imaging of patterns of cerebral blood flow (BOLD MRI) to two stimuli. These stimuli include increased carbon dioxide concentrations (causes increased cerebral blood flow) and reduced oxygen concentrations (causing decreased cerebral blood flow). In order to deliver these stimuli the investigators will use a special machine (RespiractTM) which allows for the precise control of carbon dioxide and oxygen concentrations in the lungs and blood. The precise control of carbon dioxide and oxygen in conjunction with BOLD MRI has enabled the production of detailed maps of the brain that identify areas of healthy and abnormal blood supply.

DETAILED DESCRIPTION:
OSA is associated with increased risk of cardiovascular and cerebrovascular disease compared to the general population. The mechanism for the increased stroke risk in OSA is unknown. However, the constellation of adverse pathophysiological consequences, including intermittent hypoxia and carbon-dioxide retention as a result of OSA may be detrimental to CVR and predispose the brain to ischemia. Previous studies in OSA subjects have measured CVR only using TCD. Therefore, our study will examine CVR by two methods (TCD and BOLD-MRI) with reliable and reproducible hypercapnia and independent control of oxygen saturation (RespiractTM). Patterns seen on CVR may eventually allow the identification of OSA patients who will be at greatest risk for stroke and will therefore, require aggressive risk reduction and/or treatment irrespective of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Subjects referred for sleep studies

Exclusion Criteria:

* Known cardiac, neurological or major liver or kidney disease -
* Cardioverter/defibrillator metal heart valve or pacemaker
* Vascular stent implanted within 6 weeks
* Severe claustrophobia
* Pregnancy
* Shrapnel or history of ophthalmic foreign body
* Resting oxygen saturation on room air < 95%
* Insulin-dependent diabetes
* Obstructive or restrictive lung disease such that subject is unable to walk up 2 flights of stairs
* Major depression.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community Population
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Document the diurnal differences in global CVR as measured by TCD, between those with and without OSA | Between 8pm and 7am approximately

SECONDARY OUTCOMES:
Use BOLD MRI to quantify global and regional CVR in various regions and vascular territories of the brain in subjects with OSA. | one week

CONTACTS AND LOCATIONS:
Overall Officials: Clodagh M Ryan, Principal Investigator — Toronto General Hospital
Locations (1):
- Toronto Gneral Hospital, Toronto, Ontario, Canada